CLINICAL TRIAL: NCT01095549
Title: Peripheral Artery Disease in Patients on Maintenance Hemodialysis: Risk Factors and the Effect of FIR Therapy
Brief Title: Far Infrared Therapy on Peripheral Artery Disease in Hemodialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: CHIH-CHING LIN, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V99C1-010
Record Dates: First submitted 2010-03-28; First posted 2010-03-30 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-03

CONDITIONS: Peripheral Artery Disease
Keywords: ankle-brachial index (ABI); brachial-ankle pulse wave velocity (baPWV); far infrared therapy (FIR); hemodialysis (HD); peripheral artery disease (PAD); Peripheral artery disease in hemodialysis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): HD patients who will not receive far infrared therapy in this study.
  Interventions: Device: Placebo device
- Far infrared therapy (Experimental): In this study, a WSTM TY101 FIR emitter (WS Far Infrared Medical Technology Co., Ltd., Taipei, Taiwan) will be used for FIR therapy. The electrified ceramic plates of this emitter generate electromagnetic waves with wavelengths in the range between 3 and 25 μm (a peak between 5 to 6 μm). The irradiating power density is 10 and 20 mili watt<mw>/cm2 when the top radiator is set at a distance between 30 and 20 cm above the skin surface respectively. In this study, the top radiator will be set at a height of 25 cm above the surface of bilateral lower legs and the treatment time will be set at 40 minutes for patients on maintenance HD.
  Interventions: Device: WSTM TY101 FIR emitter (Far infrared therapy)

INTERVENTIONS:
Device: WSTM TY101 FIR emitter (Far infrared therapy) — A WSTM TY101 FIR emitter (WS Far Infrared Medical Technology Co., Ltd., Taipei, Taiwan) will be used for FIR therapy. The electrified ceramic plates of this emitter generate electromagnetic waves with wavelengths in the range between 3 and 25 μm (a peak between 5 to 6 μm). The irradiating power density is 10 and 20 mili watt<mw>/cm2 when the top radiator is set at a distance between 30 and 20 cm above the skin surface respectively. In this study, the top radiator will be set at a height of 25 cm above the surface of bilateral lower legs and the treatment time will be set at 40 minutes for patients on each HD section for a year.
  Arms: Far infrared therapy
Device: Placebo device — A device without far infrared therapy
  Arms: Control group

SUMMARY:
The prevalence of peripheral artery disease (PAD) defined as ankle-brachial index (ABI) less than 0.9 was about 15~30% in patients with end stage renal disease (ESRD), which was higher than those with normal renal function. A lower ABI and a higher brachial-ankle pulse wave velocity (baPWV) are good markers to predict the risk of PAD and atherosclerosis respectively. In addition, baPWV>2,100 cm/s was shown to be related to potential PAD. ABI <0.9 was positively associated with vascular access failure in hemodialysis (HD) patients and our previous study has demonstrated that far infrared (FIR) therapy can improve access flow and unassisted patency of atrioventricular (AV) fistula.

The aims of this study are to evaluate (1) the frequency of and (2) risk factors associated with abnormal ABI and PWV as well as (3) the effect of FIR on ABI and PWV and markers related to endothelial dysfunction in HD patients.

DETAILED DESCRIPTION:
In this study, 300 HD patients will be enrolled to receive ABI and baPWV and about 90 patients (30% according to the literature review) who have abnormal ABI (<0.9) or baPWV (>2100 cm/sec) will be randomly allocated to FIR group (receiving FIR therapy for 40 minutes thrice weekly) and control group (without FIR therapy). In patients with abnormal ABI or baPWV, the effect of single or one-year treatment of FIR on the following items will be studied: (1) ABI, (2) baPWV and (3) markers related to endothelial dysfunction [including low and high density lipoprotein cholesterol (LDL and HDL), asymmetric dimethylarginine (ADMA), hypersensitive C-reactive protein (hsCRP), matrix metalloproteinase-9 (MMP-9)]. The effect of FIR on PAD or cardiovascular events during one year of follow-up will also be studied.

This study will allow us to identify the frequency of and the risk factors associated with abnormal ABI & PWV as well as the effect of single or one-year FIR therapy on ABI & PWV in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* In this study, we will include 300 patients who have received 4 hours of maintenance HD therapy three times weekly for at least 3 months

Exclusion Criteria:

* Patients with life expectancy less than 1 year
* Patients with history of active malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
ANKLE BRACHIAL INDEX | One year
  The values of the ABI were measured 10 to 30 min before HD. The ABIs will be measured by using an ABI-form device (VP1000,Colin, Komaki, Japan). The ABI will be calculated by the ratio of the ankle systolic BP divided by the arm systolic BP. The systolic BP of the arm without dialysis access and the value of the ankle systolic BP will be used for the calculation. All of the ABI and PWV will be measured twice. If the difference between them was more than 10%, a third measurement was done. The mean of the two closest values was recorded into our data base.

SECONDARY OUTCOMES:
Markers of endothelial function | One year
  Each time at the four different timings (from time 1 to time 4), we will collect blood sample 5 ml for measuring markers related to endothelial dysfunction, including low density lipoprotein cholesterol (LDL), high density lipoprotein cholesterol (HDL), asymmetric dimethylarginine (ADMA), hypersensitive C-reactive protein (hsCRP), matrix metalloproteinase-9 (MMP-9).
PAD or cardiovascular events | one year
  The effect of FIR on PAD or cardiovascular events during one year of follow-up will also be studied.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ching Lin, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan